CLINICAL TRIAL: NCT00446810
Title: Effects of a Chronical Treatment With Benfotiamine in People With Type 2 Diabetes Mellitus on Pre- and Postprandial Endothelial Function, as Well as on the Function of the Autonomic Nervous System
Brief Title: Chronic Treatment With Benfotiamine Restores Endothelial Function in People With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruhr University of Bochum (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Benfotiamine_ED_2007
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Last update posted 2007-09-27 (Estimated); Status verified 2007-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; endothelial dysfunction; benfotiamine; postprandial; autonomic neuropathy; advanced glycation end products
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — benphothiamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A1 (Active Comparator): Benfotiamine
  Interventions: Drug: Benfotiamine
- A2 (Active Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Benfotiamine
  Arms: A1
Drug: Placebo
  Arms: A2

SUMMARY:
An AGE-rich diet can induce after 2-6 weeks persistent increases in mediators linked to vascular dysfunction (e.g. TNFα, VCAM-1) in people with type 2 diabetes mellitus (T2DM). Benfotiamine (BT), the liposoluble derivative of vitamin B1, blocks several pathways common to hyperglycaemia- and AGE-induced endothelial dysfunction. We have shown that advanced glycation end products (AGE) of a regular mixed meal can acutely induce vascular dysfunction in T2DM and that this effects can be prevented by a three days pretreatment with BT.

The hypotheses of this study are that chronical treatment with benfotiamine (900 mg/day for 6 weeks) in people with type 2 diabetes mellitus:

1. prevents postprandial impairment of endothelial function after a high-AGE meal.
2. Improves fasting endothelial function.
3. Improves parameters of autonomic function in fasting and postprandial state.
4. Improves insulin sensitivity and prevents postprandial increase in insulin resistance.

DETAILED DESCRIPTION:
People with type 2 diabetes mellitus (T2DM) have a two to fivefold increase in cardiovascular mortality compared to non-diabetic controls.

Endothelial dysfunction (ED) is an early messenger of atherosclerosis and is responsible for increased vascular permeability, platelet aggregation and adhesion, leucocyte adhesion and smooth muscle cell proliferation and favours a vasoconstrictive and pro-inflammatory state.

Postprandial ED occurs not only in patients with CV disease or diabetes, but even in healthy subjects. Distinctive and cumulative effects of hyperglycemia and hypertriglyceridemia on postprandial ED have been demonstrated. Since postprandial dysmetabolism was linked to CV disease, the postprandial ED was proposed to be the mechanism connecting them. Considering that the postprandial state covers most of our daytime, interventions targeting a reduction in postprandial ED might play a decisive role in atherosclerosis prevention.

For the treatment of postprandial ED several therapeutical approaches have been suggested, such as treatment with folic acid, tetrahydrobiopterin, vitamins C and E,statins etc.

These approaches aim at reducing postprandial oxidative stress (vitamins C and E, statins and partly folic acid), postprandial hyperglycemia (insulin), postprandial hypertriglyceridemia (statins) or have a direct effect on endothelial NO production (folic acid, insulin and tetrahydrobiopterin).

Recent data suggests that advanced glycation endproducts (AGE) might also play a role in the development of ED, leading to the long-term complications of diabetes and accelerated aging. AGEs are a heterogeneous group of moieties, one of the most representative being carboxymethyllysine (CML). Diet is a major source of exogenous AGEs and the food AGE content is highly dependent on food nutrient composition, as well as on temperature, method and duration of heat application during cooking. About 10% of ingested AGEs are rapidly absorbed and partly retained into the body, where they exert different pathological effects including binding with and activation of receptors for AGE (RAGE). AGE precursors such as methylglyoxal (MG) can also activate RAGE. Endogenous MG synthesis increases in parallel with hyperglycemia in vivo. Postprandially, the absorbed and endogenously generated AGEs and MG act synergistically to decrease vascular function through direct NO scavenging or increased oxidative stress. Part of these effects can be counteracted by benfotiamine (BT), a liposoluble vitamin B1 derivative with much higher bioavailability than thiamine. BT, commonly used in the treatment of diabetic neuropathy, is a transketolase activator that directs glucose substrates to the pentose phosphate pathway. Thus, it blocks several hyperglycemia-induced pathways, one of them being endogenous AGE and dicarbonyls formation. We have recently shown that a three day pretreatment with benfotiamine can prevent postprandial ED in T2DM (Stirban et al, Diabetes Care, 2006).

This study aims at investigating the effects of a chronical treatment with benfotiamine (900 mg/day for 6 weeks) on parameters of endothelial function and autonomic neuropathy in fasting and postprandial state in people with T2DM.

We will therefore investigate 30 people with type 2 diabetes mellitus in a randomized, cross-over, double blind, placebo-controlled design. Pre- and postprandial endothelial dysfunction (flow mediated dilatation -ultrasound- and reactive hyperemia -laser-doppler-) will be investigated before and after chronical treatment with benfotiamine. Investigations will be performed in fasting state as well as 2,4 and 6 hours postprandially.

ELIGIBILITY:
Inclusion Criteria:

* People with type 2 diabetes mellitus
* Age: 30-70 years

Exclusion Criteria:

* History of myocardial infarction, stroke within the previous 6 months
* Heart failure NYHA III or more
* Malignant disease
* Severe diabetes complications
* Severe hypo- or hypertension
* Chronic alcohol abuse
* Renal failure (creatinine >2mg/dl)

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-09; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Endothelial function (flow mediated dilatation - ultrasound- and reactive hyperemia- laser doppler-) | September 2007- December 2008

SECONDARY OUTCOMES:
Parameters of autonomic neuropathy | September 2007- December 2008

CONTACTS AND LOCATIONS:
Overall Officials: Diethelm Tschoepe, Prof.PhD., Study Director — Herz- und Diabeteszentrum NRW; Alin O Stirban, PhD, Principal Investigator — Herz- und Diabeteszentrum NRW
Locations (1):
- Herz- und Diabeteszentrum NRW, Georgstr. 11, Bad Oeynhausen, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Stirban A, Negrean M, Stratmann B, Gawlowski T, Horstmann T, Gotting C, Kleesiek K, Mueller-Roesel M, Koschinsky T, Uribarri J, Vlassara H, Tschoepe D. Benfotiamine prevents macro- and microvascular endothelial dysfunction and oxidative stress following a meal rich in advanced glycation end products in individuals with type 2 diabetes. Diabetes Care. 2006 Sep;29(9):2064-71. doi: 10.2337/dc06-0531. PMID 16936154